CLINICAL TRIAL: NCT05078671
Title: Pharmacokinetic Boosting of Olaparib to Improve Exposure, Tolerance and Cost-effectiveness
Acronym: PROACTIVE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROACTIVE
Record Dates: First submitted 2021-09-22; First posted 2021-10-14 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Cancer
Keywords: olaparib; pharmacokinetic enhancement
MeSH Terms: conditions — Neoplasms | interventions — olaparib; Cobicistat

STUDY DESIGN:
Intervention Model Description: Part A: cross-over normal olaparib versus boosted olaparib. Part B: normal olaparib versus boosted olaparib in two patient groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard olaparib (Active Comparator): Olaparib 300mg twice daily
  Interventions: Drug: Olaparib
- Boosted olaparib (Experimental): Olaparib 100mg twice daily + cobicistat 150mg twice daily
  Interventions: Drug: Olaparib; Drug: Cobicistat

INTERVENTIONS:
Drug: Olaparib — olaparib treatment
Drug: Cobicistat — Pharmacokinetic booster
  Arms: Boosted olaparib

SUMMARY:
Olaparib is a poly-adenosine diphosphate ribose polymerase (PARP) inhibitor, originally used for the maintenance treatment of women with platinum-sensitive relapsed breast cancer gene (BRCA)-mutated high grade serious epithelial ovarian, fallopian tube, or peritoneal cancer, who are in response to platinum-based chemotherapy. Over the last two years, several therapeutic indications have been added to the drug label, such as first-line platinum-sensitive BRCA-mutated high grade serious epithelial ovarian, fallopian tube, or peritoneal cancer, germline BRCA1/2-mutated, human epidermal growth factor 2 (HER2-)negative, locally advanced or metastatic breast cancer and BRCA1/2-mutated metastatic castration-resistant prostate cancer, who have progressed following prior therapy. Since olaparib is very expensive, this increase of treatment population will have a significant impact on health care expenditures.

To keep healthcare affordable and accessible for all patients, innovative strategies are warranted to reduce the dose of expensive drugs, without reduction of efficacy. For olaparib, pharmacokinetic (PK) boosting can be applied. PK boosting is the lay term for administering a non-therapeutic active strong inhibitor of a metabolic enzyme, for example the cytochrome p450 enzyme 3A (CYP3A), together with a therapeutic drug that is metabolized by the same enzyme. Boosting thus increases the concentration of the therapeutic drug and allows lower doses to be administered to patients. Hence, coadministration of a reduced dose of olaparib with cobicistat, a non-therapeutic, strong inhibitor of the CYP3A can lead to equivalent exposure to olaparib. Furthermore, inhibition of CYP3A could lead to less PK variability since metabolic capacity is a prominent cause for (intra- and inter-individual) variability in systemic exposure. Predictable olaparib exposure will reduce the number of patients who are unintentionally under- or overtreated. Lastly, tumor tissue itself may express CYP3A as a detoxification or resistance mechanism. Theoretically, PK boosting may also overcome CYP3A-mediated drug resistance.

The purpose of this study is to establish the efficacy, safety and feasibility of co-administering olaparib with the PK booster cobicistat with the aim to implement boosting approach for olaparib in routine practice. The study is subdivided in two parts. In part A of the study the equivalent exposure of boosted low dose olaparib is determined compared to the normal dose. In part B of the study, non-inferiority of the boosted olaparib regimen will be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able and willing to provide written informed consent prior to screening;
* Age of 18 years or older;
* Able to measure the outcome of the study in this subject.

Part A:

* Subjects who start or are on treatment with olaparib tablets 300mg twice daily, according to the drug label and physician's discretion;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Part B:

* Subjects who start on treatment with olaparib tablets 300mg twice daily, according to the drug label and physician's discretion;
* Expected to be on olaparib treatment for ≥ 3 months;
* ECOG performance status of 0-3.

Exclusion Criteria:

* Concurrent use of other anti-cancer therapies;
* Concurrent use of potent inducers or inhibitors of the cytochrome p450 enzyme 3A3 (CYP3A4) as assessed with the Dutch drug database "G-Standaard" of the Royal Dutch Pharmacists Association(KNMP);
* Known contra-indications for treatment with cobicistat in line with the summary of product characteristics;
* Subjects with renal insufficiency defined as estimated glomerular filtration rate < 50 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Olaparib AUC0-12h | 2 weeks
  The Area-Under-the-Curve (AUC) 0-12h of olaparib.
Part B: Progression-free survival (PFS) | 12 months
  PFS is defined as time from randomization until the date of either objective radiological disease progression, or biochemical progression combined with clinical progression or death.
Part B: Dose reductions | 12 months
  Number of patients who require a dose reduction due to toxicity.

SECONDARY OUTCOMES:
Part A: Inter- and intrapatient variability of AUC0-12h | 2 weeks
  Inter- and intrapatient variability of AUC0-12h in olaparib as calculated with non-compartmental analysis.
Part A: Adverse events | 2 weeks
  Number of patients with treatment-related adverse events as assessed by CTCAE v5.0.
Part B: Health status | 12 months
  Health status as assessed with the EuroQol 5 dimensions with 5 levels questionnaire (EQ-5D-5L).
Part B: Patient satisfaction | 12 months
  Patient satisfaction as assessed with the Cancer Therapy Satisfaction Questionnaire (CTSQ).
Part B: ctDNA | 12 weeks
  Cell-free tumor nucleic acids (ctDNA) in plasma as pharmacodynamic biomarker.
Part B: Adverse events | 12 months
  Number of patients with treatment-related adverse events as assessed by CTCAE v5.0.
Part B: Productivity costs | From date of randomization until the date of end-of-treatment, assessed up to 12 months
  Productivity costs as assessed by the iMTA Productivity Costs Questionnaire (iPCQ).
Part B: Medical consumption | From date of randomization until the date of end-of-treatment, assessed up to 12 months
  Medical consumption as assessed by the iMTA Medical Consumption Questionnaire (iMCQ).

OTHER OUTCOMES:
Part A: Patient preference | 2 weeks
  Treatment preference on a 7-point Likert scale.
Part B: Intratumoral olaparib | At 8 weeks after start treatment and at the moment of progression
  Intratumoral olaparib concentration in tumor biopsy samples.

CONTACTS AND LOCATIONS:
Overall Officials: Nielka van Erp, prof. PharmD PhD, Principal Investigator — Radboud University Medical Center
Locations (10):
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Amsterdam Universitair Medische Centra, Amsterdam
  - Netherlands Cancer Institute-Antoni van Leeuwenhoek, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Universitair Medisch Centrum Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht UMC, Maastricht
  - Radboudumc, Nijmegen
  - ErasmusMC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Overbeek JK, Guchelaar NAD, Mohmaed Ali MI, Ottevanger PB, Bloemendal HJ, Koolen SLW, Mathijssen RHJ, Boere IA, Hamberg P, Huitema ADR, Sonke GS, Opdam FL, Ter Heine R, van Erp NP. Pharmacokinetic boosting of olaparib: A randomised, cross-over study (PROACTIVE-study). Eur J Cancer. 2023 Nov;194:113346. doi: 10.1016/j.ejca.2023.113346. Epub 2023 Sep 19. PMID 37806255
- [Derived] Overbeek JK, Guchelaar NAD, Mohmaed Ali MI, Sark M, Hovenier C, Kievit W, Ligtenberg MJL, Ottevanger PB, Bloemendal HJ, Koolen SLW, Mathijssen RHJ, Boere IA, Huitema ADR, Sonke GS, Opdam FL, Ter Heine R, van Erp NP. Pharmacokinetic boosting of olaparib: Study protocol of a multicentre, open-label, randomised, non-inferiority trial (PROACTIVE-B). Contemp Clin Trials Commun. 2025 Mar 29;45:101477. doi: 10.1016/j.conctc.2025.101477. eCollection 2025 Jun. PMID 40248173
- [Derived] Overbeek JK, van Erp NP, Burger DM, den Broeder AA, Koolen SLW, Huitema ADR, Ter Heine R. Population Pharmacokinetics of Cobicistat and its Effect on the Pharmacokinetics of the Anticancer Drug Olaparib. Clin Pharmacokinet. 2025 Mar;64(3):425-435. doi: 10.1007/s40262-025-01480-w. Epub 2025 Feb 5. PMID 39909979